CLINICAL TRIAL: NCT07256444
Title: Etude de faisabilité d'un Parcours de Transition à la Sortie d'Hospitalisation complète en Oncologie - Etude Pilote Monocentrique
Brief Title: Feasibility Study of a Transition Pathway at Discharge From Full Hospitalization in Oncology
Acronym: PATROL
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2023-2/AB01
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: OncoCare transition program — Interview with the coordinating nurse who reviews the patient's prescriptions and appointments, installs the electronic patient-reported outcome (ePRO) application on the patient's smartphone and explains collection of any symptoms.
  ePRO symptom monitoring by the patient on D2, D7 and D15 after discharge. The coordinating nurse phones the patient on D7 to review the symptoms reported, assess compliance with treatment and provide support. In the event of grade ≥ 2 symptoms, the nurse contacts the patient for further information and informs the referring oncologist, who decides on the course of treatment.

SUMMARY:
Patient reported outcomes (PRO) measure the health status directly reported by the patients, without external interpretation, generally collected using self-questionnaires, including online tools (ePRO). This approach is useful in early detection of signs of relapse, with reduced anxiety, improved quality of life and survival, and reduced readmissions to emergency departments in patients with advanced cancer. In the current context where hospitalization is increasingly short, the transition from hospital to home is a critical moment that poses a significant safety challenge Patient follow-up strategies help patients return home, particularly in surgery, with telephone calls from a nurse the day after or several days after discharge. In oncology, telephone calls from the pharmacist 3 days after discharge from hospital helped to identify undesirable effects of treatments. In general medicine, these calls have led to improved patient satisfaction, reduced use of emergency departments and the resolution of drug-related problems, but are costly. The introduction of post-hospitalization ePRO monitoring in oncology could ensure effective follow-up while keeping costs under control. A coordinating nurse could manage this process and play a crucial role in accompanying patients when they return home.

The study authors aimed to evaluate the feasibility of a transitional nurse consultation and ePRO follow-up on discharge from full hospitalization in oncology in this population of frail and elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* Adult patient hospitalized in an oncology unit for at least 48 hours.
* Patient capable of using a connected device, in possession of a smartphone or tablet, and with an internet connection at home.
* Patient discharged from hospital to go home.

Exclusion Criteria:

* The patient is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient considered to be at the end of life.
* Patient unable to read and understand French
* Patient discharged from hospitalization to a home care facility
* Patient having been hospitalized in a full-time inpatient setting for a scheduled procedure (chemotherapy or interventional procedure)
* Pregnant, parturient, or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients treated as inpatients in the Medical Oncology Department of Nîmes University Hospital and scheduled to be discharged and returned home.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Compliance with ePRO monitoring | Day 2
  Percentage of patients who responded to all questionnaires
Compliance with the telephone call at day 7 | Day 7
  Percentage of patients successfully contacted at day 7
Patient satisfaction with the care pathway | Day 15
  Question: "Are you satisfied with your care pathway?" (Yes/no)

SECONDARY OUTCOMES:
Quality of the transition pathway to home | Day 15
  Care Transitions Measure (CTM-3) questionnaire, where a 10-point increase reduces the risk of readmission by 14%
Quality of life as reported by the patient | Day 0
  EORTC QLQ-C30 questionnaire: The score for each subscale ranges from 0 to 100and good quality of life is associated with a high score on the functional scales and a low score on the symptom scales.
Quality of life as reported by the patient | Day 7
  EORTC QLQ-C30 questionnaire: The score for each subscale ranges from 0 to 100and good quality of life is associated with a high score on the functional scales and a low score on the symptom scales.
Quality of life as reported by the patient | Day 15
  EORTC QLQ-C30 questionnaire: The score for each subscale ranges from 0 to 100and good quality of life is associated with a high score on the functional scales and a low score on the symptom scales.
Quality of life as reported by the patient | Day 30
  EORTC QLQ-C30 questionnaire: The score for each subscale ranges from 0 to 100and good quality of life is associated with a high score on the functional scales and a low score on the symptom scales.
Patient satisfaction with their care | Day 15
  EORTC PATSAT-C33 questionnaire: The total score ranges from 0 to 100
Rate of readmissions to a healthcare facility | One month after hospitalization
  Rate of readmissions to healthcare establishments (hospitalization department, emergency room)

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Basset, Principal Investigator — CHU de Nimes
Locations (1):
- Centre Hospitalier de Nimes, Nîmes, France